CLINICAL TRIAL: NCT00041405
Title: Mechanisms of Pro-Thrombosis in Diabetes Mellitus -- Ancillary to BARI 2D
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1179; R01HL069146 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2002-07-09 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Non-insulin Dependent; Coronary Disease; Thrombosis; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Diabetes Mellitus, Type 2; Coronary Disease; Thrombosis; Diabetes Mellitus

SUMMARY:
To determine the effect of the method of hyperglycemic management on pro- thrombotic potential in diabetic subjects.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease is the leading cause of death in patients with diabetes. The BARI 2D study is designed to determine the potential value of specific treatment regimens for those with diabetes and will test the hypothesis that "with a target HbA1C of less than 7.5%, a strategy of hyperglycemic management directed at insulin sensitization results in lower 5 year mortality compared to a strategy of insulin provision." This ancillary study is designed to provide mechanistic insight into potential benefits derived from two different treatment strategies employed by characterizing the thrombotic potential in those patients assigned to the aggressive medical management strategy and long-range goal is to demonstrate that treatment of diabetes with regimens that reduce thrombotic potential decreases cardiovascular risk. The results of this ancillary study should help to define the extent to which specific regimens diminish the pro-thrombotic state.

The study is in response to an initiative on Ancillary Studies in Heart, Lung, and Blood Disease Trials released in June, 2000.

DESIGN NARRATIVE:

Thrombotic potential will be assessed by determination of both platelet reactivity and thrombin generation and activity. Preliminary studies have found that patients with diabetes have increased coronary intervention. Further, thrombin generation and activity is increased in diabetic subjects. Preliminary evidence suggests that treatment with an insulin-sensitizing regimen reduces platelet reactivity, thrombin generation and thrombin activity. The BARI 2D study is ideally suited for determination of the effect of the method of glycemic control on pro-thrombotic potential. In aim 1 the investigators will determine platelet reactivity before and during the first year of treatment in patients randomized to medical treatment and randomized also to either an insulin-sensitizing regimen or an insulin-providing regimen. They will use a flow cytometry-based assay of platelet function that they have developed and validated. In aim 2 they will determine the effect of treatment on thrombin generation and activity in the same group of patients. Thrombin generation will be determined by measuring the concentration in blood of a cleavage fragment (prothrombin fragment 1+2). Thrombin activity will be determined by measuring the concentration in blood of a second cleavage fragment (fibrinopeptide A). The results of the studies will determine the effect of the method of hyperglycemic management on pro-thrombotic potential. Further, these results will define the importance of prothrombotic potential in diabetic subjects while potentially identifying new therapeutic targets in patients with diabetes and other insulin resistant states.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-07; Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schneider — University of Vermont & State Agricultural College

REFERENCES:
- [Background] Keating FK, Sobel BE, Schneider DJ. Effects of increased concentrations of glucose on platelet reactivity in healthy subjects and in patients with and without diabetes mellitus. Am J Cardiol. 2003 Dec 1;92(11):1362-5. doi: 10.1016/j.amjcard.2003.08.033. PMID 14636925